CLINICAL TRIAL: NCT01294306
Title: Phase II Trial of the Akt Inhibitor MK-2206 Plus Erlotinib (OSI-774) in Patients With Advanced Non-small Cell Lung Cancer Who Have Progressed After Previous Response (Including Stable Disease) With Erlotinib Therapy
Brief Title: MK2206 and Erlotinib Hydrochloride in Treating Patients With Advanced Non-Small Cell Lung Cancer Who Have Progressed After Previous Response to Erlotinib Hydrochloride Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02578; NCI-2011-02578 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000695056; CHNMC-PHII-108; PhII-108 (Other: City of Hope Comprehensive Cancer Center); 8698 (Other: CTEP); N01CM00038 (NIH); N01CM00071 (NIH); N01CM62209 (NIH); P30CA033572 (NIH)
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Adenosquamous Lung Carcinoma; Bronchioloalveolar Carcinoma; Large Cell Lung Carcinoma; Lung Adenocarcinoma; Recurrent Non-Small Cell Lung Carcinoma; Squamous Cell Lung Carcinoma
MeSH Terms: conditions — Adenocarcinoma, Bronchiolo-Alveolar; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — MK 2206; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Akt inhibitor MK2206, erlotinib hydrochloride) (Experimental): Patients receive Akt inhibitor MK2206 PO QOD of a 28-day course, and erlotinib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor MK2206; Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK2206
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies the side effects and how well Akt inhibitor MK2206 (MK2206) and erlotinib hydrochloride works in treating patients with advanced non-small cell lung cancer who have progressed after previous response to erlotinib hydrochloride therapy. MK2206 and erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy (with the primary endpoint of disease control at 12 weeks) and tolerability of the combination of MK2206 plus erlotinib (erlotinib hydrochloride) in previously erlotinib-treated patients with recurrent or progressive advanced non-small cell lung cancer (NSCLC) whose tumors are either epidermal growth factor receptor (EGFR) mutated or EGFR wild-type.

SECONDARY OBJECTIVES:

I. To determine progression-free survival of previously erlotinib-treated patients with NSCLC who are treated with MK2206 plus erlotinib. II. To determine the overall survival of previously erlotinib-treated patients with NSCLC who are treated with MK2206 plus erlotinib.

III. To assess the toxicity experienced by previously erlotinib-treated patients with NSCLC treated with MK2206 plus erlotinib. IV. To perform correlative analysis of tumor biomarkers to assess, in a preliminary manner, the association between tumor mutations and/or abnormalities and clinical outcome of previously erlotinib-treated patients with NSCLC treated with MK2206 plus erlotinib.

OUTLINE:

Patients receive Akt inhibitor MK2206 orally (PO) every other day (QOD) of a 28-day course, and erlotinib hydrochloride PO once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 12 weeks for one year and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed non-small cell lung cancer of any histologic subtype

  * NOTE: epidermal growth factor receptor (EGFR) mutational status (either wild-type or positive for an activating mutation) will be determined for all patients on this study; commercial assays for EGFR mutation status are allowed; knowledge of EGFR mutational status is not required at the time of protocol entry but should be determined or known before the end of course 2; however, if one of the strata is temporarily closed to accrual, knowledge of EGFR mutational status will be required prior to protocol entry
* Patients may have measurable or non-measurable disease; x-rays and/or scans for disease assessment of measurable disease must have been completed within 28 days prior to registration
* Patients must have radiologic or clinical progressive disease following prior benefit (response or stable disease) to EGFR-tyrosine kinase inhibitor (TKI) therapy (e.g., erlotinib) administered either as a single agent or in combination with other agents for at least 12 weeks prior to progression; Note: patients may have received intervening systemic therapy after EGFR-TKI progression); additionally, patients must have documentation of radiographic progression within the preceding three months prior to study entry
* Prior cytotoxic chemotherapy is allowed; any number of prior chemotherapy regimens is also allowed; prior cetuximab therapy is also allowed; NOTE: a patient with an EGFR activating mutation who has received EGFR-TKI therapy as first line therapy, but has not received platinum-based chemotherapy, would be considered eligible for this trial
* Karnofsky performance status >= 60%
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelet count >= 100,000/mcL
* Total bilirubin =< upper institutional normal limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine =< upper institutional normal limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Prior to the first patient registration, this study must be institutional review board approved; a copy of the institutional review board (IRB) approval for each site involved must be given to the Data Coordinating Center at City of Hope
* Women of childbearing potential and men must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treating physician immediately
* Patients on coumadin should have their international normalized ratio (INR) monitored at least once per week or more frequently depending on the investigator's judgment; there have been some case reports of increased INR when coumadin is co-administered with erlotinib
* Ability to understand and the willingness to sign a written informed consent document
* Patients should have tumor tissue (either fresh frozen tumor tissue or paraffin-embedded tumor tissue) available for retrieval; if an endobronchial lesion is present or suspected, bronchoscopy is recommended as a source of fresh tissue; tissue blocks or unstained slides from the time of original diagnosis are acceptable if repeat biopsy is not feasible

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have any ongoing grade 2 or greater toxicity from a prior treatment
* Patients may not be receiving any other investigational agents
* Patients with symptomatic brain metastases should be excluded from this clinical trial; patients with asymptomatic controlled or treated (e.g., with radiation and/or surgery) brain metastases are otherwise eligible as long as corticosteroids given expressly for brain metastases (mets) have been stopped for at least 14 days
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206 or erlotinib
* Caution must be observed for patients receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP 450 3A4); although these patients are still potentially eligible, close monitoring is required for toxicity
* Preclinical studies demonstrated the potential of MK-2206 for induction of hyperglycemia in all preclinical species tested; patients with diabetes or in risk for hyperglycemia should not be excluded from trials with MK-2206, but the hyperglycemia should be well controlled on oral agents before the patient enters the trial
* Preclinical studies indicated transient changes in corrected QT (QTc) interval during MK-2206 treatment; prolongation of QTc interval is potentially a safety concern while on MK-2206 therapy; cardiovascular: baseline Fridericia QT (QTcF) > 450 msec (male) or QTcF > 470 msec (female) will exclude patients from entry on study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with this combination
* Human immunodeficiency (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Prior MK-2206 therapy is not allowed
* Patients unable to swallow MK-2206 tablets and erlotinib tables whole are ineligible; (the tablets cannot be crushed or broken)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo Lara, Principal Investigator — University of California, Davis
Locations (7):
- United States (7):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- EGFR-Mutated Tumors: Patients with EGFR-mutated tumors.
- EGFR Wild-Type Tumors: Patients with EGFR wild-type tumors.
Period: Overall Study
Arm/Group | EGFR-Mutated Tumors | EGFR Wild-Type Tumors
Started | 45 | 35
Completed | 45 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EGFR-Mutated Tumors | EGFR Wild-Type Tumors | Total
Number analyzed (Participants) | 45 | 35 | 80
Age, Continuous [Median (Full Range); unit: years] | 64 [44 to 86] | 63 [40 to 83] | 64 [40 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 20 | 51
  Male | 14 | 15 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 6 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 20 | 27 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 45 | 35 | 80

OUTCOME MEASURES:

1. Primary Outcome: Disease-control Rate
Description: Disease-control rate defined as response rate + stable disease at 12 weeks. Stable disease must have been achieved for 12 weeks or longer. Response evaluated per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
Time Frame: At 12 weeks
Measure: Number; unit: percentage of subjects
Arm/Group | EGFR-Mutated Tumors | EGFR Wild-Type Tumors
Number analyzed (Participants) | 45 | 35
percentage of subjects | 40 | 43

2. Primary Outcome: Objective Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response = CR + PR
Time Frame: Up to 2 years
Measure: Number; unit: percentage of subjects
Arm/Group | EGFR-Mutated Tumors | EGFR Wild-Type Tumors
Number analyzed (Participants) | 45 | 35
percentage of subjects | 9 | 3

3. Secondary Outcome: Median Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EGFR-Mutated Tumors | EGFR Wild-Type Tumors
Number analyzed (Participants) | 45 | 35
Months | 4.4 [2.7 to 6.6] | 4.6 [2.9 to 8.5]

4. Secondary Outcome: Toxicity of Akt Inhibitor MK2206 Plus Erlotinib Hydrochloride
Description: Toxicities of Grade 3 or higher Attributed to Akt inhibitor MK2206 plus erlotinib hydrochloride, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | EGFR-Mutated Tumors | EGFR Wild-Type Tumors
Number analyzed (Participants) | 45 | 35
participants
  Anemia | 0 | 1
  Diarrhea | 5 | 5
  Mucositis | 4 | 1
  Nausea | 1 | 2
  Vomiting | 0 | 1
  Fatigue | 5 | 3
  Skin infection | 0 | 1
  Lung infection | 2 | 0
  Urinary tract infection | 1 | 1
  Creatinine increased | 0 | 1
  Lymphocyte count decreased | 6 | 3
  Anorexia | 0 | 1
  Dehydration | 3 | 0
  Hyperglycemia | 3 | 0
  Hypokalemia | 2 | 0
  Hyponatremia | 0 | 2
  Hypophophatemia | 1 | 0
  Myalgia | 1 | 0
  Neoplasm | 0 | 1
  Dyspnea | 1 | 1
  Dry skin | 0 | 3
  Erythema multiforme | 1 | 0
  Skin peeling (feet) | 0 | 1
  Pruritus | 0 | 1
  Rash | 9 | 3
  Hypertension | 1 | 0

5. Secondary Outcome: Median Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Event defined as death due to any cause.
Time Frame: Up to 2 Years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EGFR-Mutated Tumors | EGFR Wild-Type Tumors
Number analyzed (Participants) | 45 | 35
Months | 10.6 [8.6 to 23.2] | 11.1 [7.3 to 22.1]

ADVERSE EVENTS:
Time Frame: Adverse events collected over a period of 4 years and 8 months.
Description: Includes all adverse events regardless of attribution and grade.
Arm/Group | EGFR-Mutated Tumors | EGFR Wild-Type Tumors
Serious Adverse Events (participants affected / at risk) | 17/45 | 21/35
Other Adverse Events (participants affected / at risk) | 45/45 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EGFR-Mutated Tumors (N=45) | EGFR Wild-Type Tumors (N=35)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 7 (9) | 3 (3)
Death NOS (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 3 (3) | 3 (3)
Paronychia (Infections and infestations) | 1 (1) | 1 (2)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 5 (8) | 6 (8)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Progressive Disease, Death NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrown hair (eyelashes) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
skin discoloration (green, gray) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EGFR-Mutated Tumors (N=45) | EGFR Wild-Type Tumors (N=35)
Anemia (Blood and lymphatic system disorders) | 17 (46) | 19 (79)
Aortic Aneurysm (Blood and lymphatic system disorders) | 0 (0) | 1 (8)
Aortic aneurysm (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ascending aortic aneurysm (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (2)
Heart failure (Cardiac disorders) | 0 (0) | 1 (2)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 2 (4)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (5)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
fluid in ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (3) | 1 (1)
Blurry Vision (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (3)
Conjunctivitis (Eye disorders) | 3 (5) | 0 (0)
Dry eye (Eye disorders) | 8 (33) | 3 (8)
Eye pain (Eye disorders) | 1 (1) | 1 (2)
Ingrown eyelashes (Eye disorders) | 0 (0) | 1 (2)
Redness Irritation (Eye disorders) | 1 (1) | 0 (0)
Sensitivity to sun (Eye disorders) | 0 (0) | 1 (1)
Watery Eyes (Eye disorders) | 1 (1) | 0 (0)
eye irritation (Eye disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 7 (11) | 6 (17)
Bloating (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (21) | 10 (35)
Diarrhea (Gastrointestinal disorders) | 36 (123) | 27 (114)
Dry mouth (Gastrointestinal disorders) | 9 (21) | 5 (7)
Dyspepsia (Gastrointestinal disorders) | 3 (5) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (5) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (3) | 2 (3)
Gastritis (Gastrointestinal disorders) | 2 (11) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (8) | 3 (5)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (2) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 2 (5) | 1 (3)
Intermittent stomach aches (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 22 (44) | 10 (21)
Nausea (Gastrointestinal disorders) | 12 (25) | 14 (26)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (3)
Oral pain (Gastrointestinal disorders) | 2 (2) | 2 (5)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (3) | 2 (2)
Stomach Flu (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 10 (14) | 8 (10)
rough in mouth/sips (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 4 (5) | 6 (6)
Death NOS (General disorders) | 11 (11) | 10 (10)
Edema face (General disorders) | 0 (0) | 1 (2)
Edema limbs (General disorders) | 7 (11) | 6 (12)
Fatigue (General disorders) | 35 (115) | 30 (101)
Fever (General disorders) | 5 (7) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0)
Neck edema (General disorders) | 1 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (10) | 4 (16)
Pain (General disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (2) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (3)
Infected abrasion (Infections and infestations) | 0 (0) | 1 (1)
Infected abrasion wound (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (4) | 1 (1)
Nail infection (Infections and infestations) | 1 (5) | 1 (14)
Otitis externa (Infections and infestations) | 0 (0) | 1 (2)
Otitis media (Infections and infestations) | 1 (2) | 1 (3)
Paronychia (Infections and infestations) | 9 (20) | 5 (25)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Sinus (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (3) | 2 (7)
Skin infection (Infections and infestations) | 0 (0) | 2 (5)
Upper respiratory infection (Infections and infestations) | 2 (2) | 4 (8)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (5)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (2)
Vulval infection (Infections and infestations) | 1 (3) | 0 (0)
Yeast Infection (Infections and infestations) | 1 (1) | 0 (0)
oral thrush (Infections and infestations) | 0 (0) | 1 (2)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (5)
Activated partial thromboplastin time pr (Investigations) | 2 (2) | 1 (13)
Alanine aminotransferase increased (Investigations) | 7 (10) | 5 (17)
Alkaline phosphatase increased (Investigations) | 14 (34) | 7 (20)
Aspartate aminotransferase increased (Investigations) | 11 (21) | 9 (43)
Blood bilirubin increased (Investigations) | 13 (39) | 6 (23)
Cholesterol high (Investigations) | 1 (3) | 1 (6)
Creatinine increased (Investigations) | 7 (34) | 12 (75)
INR increased (Investigations) | 2 (2) | 2 (39)
Lymphocyte count decreased (Investigations) | 14 (46) | 15 (56)
Neutrophil count decreased (Investigations) | 3 (7) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (2)
Right bundle branch block (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 11 (35) | 13 (71)
White blood cell decreased (Investigations) | 7 (35) | 4 (8)
Anorexia (Metabolism and nutrition disorders) | 23 (47) | 21 (53)
Dehydration (Metabolism and nutrition disorders) | 3 (5) | 4 (4)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (54) | 12 (26)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (9)
Hypernatremia (Metabolism and nutrition disorders) | 4 (9) | 3 (6)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 16 (28) | 10 (66)
Hypocalcemia (Metabolism and nutrition disorders) | 8 (24) | 8 (14)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (22) | 5 (10)
Hypokalemia (Metabolism and nutrition disorders) | 8 (16) | 5 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 3 (8)
Hyponatremia (Metabolism and nutrition disorders) | 12 (21) | 11 (13)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (15) | 5 (10)
LDH Increased (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 5 (25) | 5 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (10) | 2 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (25) | 8 (16)
Back spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (18) | 5 (9)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4 (12) | 1 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (10)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (8)
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (4)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (19) | 4 (11)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7) | 4 (9)
hand cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
leg cramps (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 (22) | 20 (20)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 3 (11) | 1 (11)
Dizziness (Nervous system disorders) | 6 (10) | 4 (6)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 16 (48) | 11 (27)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (14) | 4 (8)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (2) | 4 (13)
Paresthesia (Nervous system disorders) | 2 (9) | 4 (8)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (14) | 4 (25)
sciatic like pain (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 3 (12) | 2 (3)
Confusion (Psychiatric disorders) | 4 (5) | 1 (1)
Crying spells (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (11) | 3 (5)
Hallucinations (Psychiatric disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (20) | 3 (11)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (17)
Hematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (6)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (2)
Vaginal dryness (Reproductive system and breast disorders) | 1 (2) | 1 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (20) | 5 (10)
Blood Streaked Sputum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest congestion, possible infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (66) | 14 (67)
Diminished Breath Sounds (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (34) | 15 (35)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 4 (10)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 1 (4)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (8)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory illness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (9) | 4 (5)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 3 (10)
chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
chest tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (11) | 5 (26)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Cracked skin on feet (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decadron rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Desquamation of lips (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Desquamation right palm/fingers (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 26 (119) | 24 (115)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 5 (17) | 3 (4)
Erythematous scaly rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Finger Cracks (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Finger tip cracks (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Hand Food Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (9)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 2 (5) | 1 (3)
In grown toenail (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Ingrown toe nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrown toe nail - right foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrown toenail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Mottle rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (5)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (30)
Palmar-plantar erythrodysesthesia syndro (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Peeling @ bottoms of feet (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Peeling @bottoms of feet (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 16 (59) | 15 (39)
Rash acneiform (Skin and subcutaneous tissue disorders) | 22 (80) | 13 (54)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 23 (92) | 17 (86)
Scaling on toes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (8) | 2 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (5) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
cracks on feet (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
decadron rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
desquamation of palm/fingers (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
desquamation of r palm/fingers (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
desquamation, right palm/fingers (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
dry desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
finger cracks (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
finger tip cracks (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (6)
ingrown toenail (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
scaling on toes (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
skin cracks (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
subcutaneous lesion in elbow (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 17 (85) | 12 (45)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less